CLINICAL TRIAL: NCT07325201
Title: Mitigating Diabetic Ketoacidosis in People With T1D and Chronic Kidney Disease on an SGLT1&2 Inhibitor: Ketosis Risk Factor Determination and Incorporation Into an Enhanced Glucose Ketone Report
Brief Title: Reducing Risk of Diabetic Ketoacidosis in Type 1 Diabetes and Kidney Disease Using Continuous Ketone Monitoring
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-153; 1U01DK143379 (NIH)
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus; Chronic Kidney Disease (CKD) With Diabetes Mellitus (DM); Chronic Kidney Disease
Keywords: Type 1 Diabetes; Chronic Kidney Disease; Continuous Glucose Monitoring; Diabetic Ketoacidosis; Continuous Ketone Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Renal Insufficiency, Chronic; Diabetic Ketoacidosis

STUDY DESIGN:
Intervention Model Description: All patients will be started on sotagliflozin at a dose of 200 mg/d. After 3 months of sotagliflozin 200 mg/d, patients who do not achieve good glycemic control (Time In Range >60%) and who have moderate or no chronic kidney disease (estimated Glomerular Filtration Rate >60) will be offered the option to increase sotagliflozin to 400 mg/d. The decision to increase sotagliflozin dose will be a shared decision between the study subject and the study investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotagliflozin (Experimental): In this single arm trial, all patients will be started on sotagliflozin at a dose of 200mg/d. After 3 months of sotagliflozin 200 mg/d, patients who do not achieve good glycemic control (TIR >60%) and who have moderate or no CKD (eGFR >60) will be offered the option to increase sotagliflozin to 400mg/d. All other participants will continue taking 200 mg sotagliflozin daily.
  Interventions: Drug: Sotagliflozin initiation

INTERVENTIONS:
Drug: Sotagliflozin initiation — All patients will be started on sotagliflozin at a dose of 200mg/d. After 3 months of sotagliflozin 200 mg/d, patients who do not achieve good glycemic control (TIR >60%) and who have moderate or no CKD (eGFR >60) will be offered the option to increase sotagliflozin to 400mg/d. The decision to increase sotagliflozin dose will be a shared decision between the study subject and the study investigators. All other participants will continue taking 200 mg sotagliflozin daily. After completing all study visits, all participants will stop taking sotagliflozin and continue care with their healthcare provider(s).

SUMMARY:
The goal of this clinical trial is to develop and evaluate a novel diabetes ketoacidosis risk mitigation strategy to support the safe use of sodium-glucose cotransporter-2 inhibitors (SGLT2i) therapy in participants with type 1 diabetes (T1D) and mild to moderate chronic kidney disease (CKD). The main objectives of this study are to:

1. Evaluate how ketone metrics differ between participants with mild to moderate chronic kidney disease and those with normal renal function in three time periods.
2. Identify potentially modifiable ketosis risk factors.
3. Use continuous glucose monitoring (CGM) and continuous ketone monitoring (CKM) data prior to and following treatment to determine ketosis risk factors and gain knowledge to further refine reporting of risk factors.
4. Gather information on how participants and clinicians like and use the CGM/CKM reports.

Participants will be asked to:

* Meet with study investigators to determine if they are eligible
* Sign written informed consent
* Take a pregnancy test, if applicable
* Have blood taken to assess kidney function and hemoglobin A1c
* Take the study medication, following the study team instructions
* Wear the study provided sensor throughout participation.
* Complete 5 in person visits, and 11 phone check ins over a nine-month period
* Provide feedback on the usefulness of CGM/CKM reports

DETAILED DESCRIPTION:
It is estimated that 1.8 million people in the U.S. have type 1 diabetes (T1D) and of these, at least 20% have chronic kidney disease (CKD). Sodium-glucose cotransporter inhibitors (SGLT2i) and similar medications improve glycemic control and are cardioprotective and kidney protective. However, in trials of SGLT2i as an adjunct to insulin in patients with T1D, potential benefits were not fully realized due to increased incidence of diabetic ketoacidosis (DKA). Future approval of SGLT2i for T1D will depend on a more comprehensive understanding of ketosis risks and feasible strategies for prevention of DKA. Use of continuous ketone monitoring (CKM) may allow for the safe use of SGLT2i in patients with T1D, but patient use of the ketone data in real-time and patient and provider use of a retrospective combined CGM/CKM report will both be critical components of how CKM data may help facilitate the safe use of SGLT2i therapy to improve health outcomes.

The overall goals of this study are to develop and evaluate a novel DKA risk mitigation strategy to support the safe use of SGLT2i therapy in patients with T1D. The investigators propose studying SGLT2i medications with a focus on patients with T1D and mild to moderate CKD; this group is the most likely to benefit from the SGLT2i kidney protective effects and, once approved for use in T1D, patients at risk for kidney disease may be prioritized for treatment with SGLT2i therapy. The DKA risk mitigation strategy will leverage early detection of risk for DKA through CKM technology and our team's expertise in developing and implementing standardized, comprehensive, and clinically relevant reports for CGM data. The combined CGM/CKM report, in addition to continuous glucose and ketone data, will incorporate patient data on potentially modifiable ketosis risk factors. The CGM/CKM report will be refined taking into account the preferences of patients and providers, ensuring an accessible and interpretable user interface and supporting sustained behavior changes to prevent episodes of ketosis and to ensure that when episodes of ketosis do occur, they do not progress to DKA. This study builds on our extensive clinical and research expertise in diabetes care, qualitative and quantitative analyses, and leadership in optimization of CGM reports to improve glycemic control and long-term clinical outcomes while preventing DKA in patients with T1D and CKD progression.

The medication to be used in this study is sotagliflozin, a combination SGLT 1 and 2 inhibitor manufactured by Lexicon Pharmaceuticals (The Woodlands, TX). The medication is approved by FDA in the United States as treatment for heart failure, including for those with T2D. Sotagliflozin is administered orally in the outpatient setting. It has also been approved in Europe by the European Medicines Agency as an adjunct to insulin therapy to improve glycemic control in adults with T1D with a BMI >27 kg/m2, who have not achieved adequate glycemic control despite optimal insulin therapy. The drug is sold in the United States as Zynquista and is currently available for prescription use through regular pharmacy channels. The decision to increase sotagliflozin dose will be a shared decision between the study subject and the study investigators.

The study device used is the combined continuous glucose and ketone monitor (CGKM) manufactured by Abbott Diabetes (Chicago, IL). The device uses a sensor placed subcutaneously to measure interstitial fluid levels of glucose and BHB every 1 minute and via the attached transmitter on the skin surface, transmit the data to a receiver (or smartphone application). The device is currently pending FDA approval; investigators will ensure the device is FDA approved prior to beginning any study-related activities.

Patients will receive real-time alerts from the device at the manufacturer's programed ketone thresholds (to be determined per the commercially available CKM device). Patients will also be educated on proper identification and management of acute ketonemia, including how to use the data from the CKM in real-time to recognize and treat ketone levels as soon as they arise. This will be based on our own internal standing orders for "Adult Diabetes Management: Hyperglycemia and Ketoacidosis" which is based upon the ADA guidance for hyperglycemia management as well as informed by the STOP protocol to guide CHO intake along with appropriate insulin dosing. This standing order will provide guidance for fluids, insulin, and CHO intake based on the glucose and ketone levels, and factor into account presence and severity of symptoms in when to recommend seeking care in an emergency department. The CKM will have novel trend arrows about ketosis which will also be incorporated into the real-time ketone management guidance (e.g. increase insulin bolus 10% if trend arrows are pointing up). Patients will be provided with detailed instructions as well as a paper wallet card to always carry with them.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Males and females; Ages 18-75.
* Diagnosis of type 1 diabetes, based on a clinical diagnosis with onset at least 3 months prior to screening.
* Using an automated insulin delivery system (AID) or multiple daily injections (MDI), (defined by use of rapid analogue with meals and approved long-acting analogue (e.g. detemir or glargine)).
* Most recent eGFR ≥30 (and within prior 12 months).
* HbA1c <10%. 8) Have had ≥1 primary or specialty ambulatory visit(s) in the past year in the HealthPartners care system.
* Have never been prescribed SGLT2i medications.
* Must be willing and able to wear a CGM/CKM device and willing to follow the study protocol.
* Must be able to read and speak English.
* Use of adequate contraception for the duration of the study be the women of childbearing potential.
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone, internet access).

Exclusion Criteria:

* Pregnancy, lactation, planning to become pregnant or unwillingness to be on contraception during the trial.
* Any form of diabetes other than T1D.
* Any history of use of sodium-glucose cotransporter inhibitors and use of other non-insulin glucose lowering medication within the last 6 months.
* Chronic systemic corticosteroids (>4 consecutive weeks) within 6 months before screening or planned use during the study period.
* History of diabetic ketoacidosis within 3 months of screening or 2 or more episodes of DKA within the last year.
* History of multiple (≥ 3 infections) genital mycotic infections within 6 months of screening.
* Hypotension at screening as defined as, systolic blood pressure < 90 and diastolic blood pressure < 60 with symptoms of low blood pressure (confusion, dizziness, lightheadedness, fainting, heart palpitations).
* History of a level 3 hypoglycemic event (as defined by ADA criteria) within 3 months of screening.
* Recent myocardial infarction, stroke, hospitalization for unstable angina or heart failure within 3 months prior to screening.
* New York Heart Association Class IV heart failure.
* CKD-EPI estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2.
* Impairment of systems and organs that may increase their risk of participating in the intervention study or compromise the results (for example: end stage kidney disease, active liver dysfunction, gastroparesis, anemia, organ transplant).
* Active Hepatitis B or C, or tuberculosis.
* Abnormal liver function at screening defined as any of the following: aspartate aminotransferase (AST) >2X upper limit of the normal reference range (ULN), ALT >2X ULN, serum total bilirubin (TB) >1.5X ULN.
* History of severe acquired immune deficiency syndrome or human immunodeficiency virus (HIV) infection or severely immunocompromised status, in the opinion of the investigator, including, but not limited to patients who have undergone organ or bone marrow transplantation. HIV positive patients who are on stable immunosuppressive therapy and have undetectable viral load may be eligible for inclusion in the study, subject to the investigator's discretion.
* Current or past history of decompensated cirrhosis (defined as variceal bleeding, ascites or hepatic encephalopathy), and/or known diagnosis of cirrhosis.
* Cancer treatment (excluding non-melanoma skin cancer treated by excision, carcinoma in situ of the cervix or uterus, ductal breast cancer in situ, resected non-metastatic breast or prostate cancer) within one year of screening.
* History of kidney transplant.
* CKD from a known cause other than T1D.
* A diagnosed eating disorder.
* BMI <22.
* Adherence to a very low CHO or ketogenic diet.
* A foot amputation.
* Non-healing wounds of extremities.
* Inability to perform the study follow up/ unwilling to wear the investigational device.
* Heavy alcohol use (for men, ≥5 drinks on any day or ≥15 drinks per week; for women, ≥4 drinks on any day or ≥8 drinks per week) at screening, history of alcohol use disorder or binge drinking.
* Participation in another treatment or intervention study within the past six weeks.
* Any condition or factor that would compromise the participant's safety or conduct of the study (for example: cognitive impairment, bipolar disorder, or eating disorder) or any other reason the PI deems that the patient should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in % time in ketone range >1.5/mmol/L | Baseline 3 months to 3 months following sotagliflozin initiation
Number of episodes of diabetic ketoacidosis | 3 months following sotagliflozin initiation
  ADA/EASD consensus on hyperglycemia definition of DKA will be used for the definition of DKA (must meet all 3 criteria: Glucose ≥200 mg/dL (11.1 mmol/L) OR prior history of diabetes; BHB concentration ≥3.0 mmol/L OR urine ketone strip 2+ or greater; pH <7.3 and/or bicarbonate concentration <18 mmol/L)

SECONDARY OUTCOMES:
Change in mean ketone level | Baseline 3 months to 3 months following sotagliflozin initiation
Highest ketone level observed | 3 months following sotagliflozin initiation
Number of episodes of ketosis with >=15 minutes at >1.5 mmol/L | 3 months following sotagliflozin initiation
Number of prolonged episodes of ketosis with >=120 minutes at >1.5 mmol/L | 3 months following sotagliflozin initiation
Change in % time in ketone range >=3.0/mmol/L | Baseline 3 months to 3 months following sotagliflozin initiation
Change in mean ketone level | Baseline 3 months to 3 months following sotagliflozin titration
  After 3 months of sotagliflozin 200 mg/d, participants with poor glycemic control and mild to no chronic kidney disease will switch to sotagliflozin 400 mg/d, with shared decision making
Highest ketone level observed | 3 months following sotagliflozin titration
  After 3 months of sotagliflozin 200 mg/d, participants with poor glycemic control and mild to no chronic kidney disease will switch to sotagliflozin 400 mg/d, with shared decision making
Number of episodes of ketosis with >=15 minutes at >1.5 mmol/L | 3 months following sotagliflozin titration
  After 3 months of sotagliflozin 200 mg/d, participants with poor glycemic control and mild to no chronic kidney disease will switch to sotagliflozin 400 mg/d, with shared decision making
Number of prolonged episodes of ketosis with >=120 minutes at >1.5 mmol/L | 3 months following sotagliflozin titration
  After 3 months of sotagliflozin 200 mg/d, participants with poor glycemic control and mild to no chronic kidney disease will switch to sotagliflozin 400 mg/d, with shared decision making
Change in % time in ketone range >=3.0/mmol/L | Baseline 3 months to 3 months following sotagliflozin titration
  After 3 months of sotagliflozin 200 mg/d, participants with poor glycemic control and mild to no chronic kidney disease will switch to sotagliflozin 400 mg/d, with shared decision making

OTHER OUTCOMES:
Change in A1c | 3- and 6-months following sotagliflozin initiation and titration
Change in CGM metrics | 3-and 6-months following sotagliflozin initiation and titration
Reduction in insulin total daily dose | 3-and 6-months following sotagliflozin initiation and titration

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bergenstal, MD, Principal Investigator — HealthPartners/Park Nicollet International Diabetes Center
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Steering committee will agree upon a publication and NIH Public Access Policy

REFERENCES:
- [Background] Bergenstal RM. Continuous glucose monitoring: transforming diabetes management step by step. Lancet. 2018 Apr 7;391(10128):1334-1336. doi: 10.1016/S0140-6736(18)30290-3. Epub 2018 Feb 16. No abstract available. PMID 29459022
- [Background] Maines E, Pertile R, Cauvin V, Soffiati M, Franceschi R. Glucose metrics improvement in youths with type 1 diabetes using the Ambulatory Glucose Profile report: A real-world study. Diabetes Res Clin Pract. 2024 Jun;212:111720. doi: 10.1016/j.diabres.2024.111720. Epub 2024 May 24. PMID 38797262
- [Background] Huang J, Yeung AM, Bergenstal RM, Castorino K, Cengiz E, Dhatariya K, Niu I, Sherr JL, Umpierrez GE, Klonoff DC. Update on Measuring Ketones. J Diabetes Sci Technol. 2024 May;18(3):714-726. doi: 10.1177/19322968231152236. Epub 2023 Feb 16. PMID 36794812
- [Background] Goldenberg RM, Gilbert JD, Hramiak IM, Woo VC, Zinman B. Sodium-glucose co-transporter inhibitors, their role in type 1 diabetes treatment and a risk mitigation strategy for preventing diabetic ketoacidosis: The STOP DKA Protocol. Diabetes Obes Metab. 2019 Oct;21(10):2192-2202. doi: 10.1111/dom.13811. Epub 2019 Jun 30. PMID 31183975
- [Background] Garg SK, Peters AL, Buse JB, Danne T. Strategy for Mitigating DKA Risk in Patients with Type 1 Diabetes on Adjunctive Treatment with SGLT Inhibitors: A STICH Protocol. Diabetes Technol Ther. 2018 Sep;20(9):571-575. doi: 10.1089/dia.2018.0246. Epub 2018 Aug 21. No abstract available. PMID 30129772
- [Background] Chow E, Clement S, Garg R. Euglycemic diabetic ketoacidosis in the era of SGLT-2 inhibitors. BMJ Open Diabetes Res Care. 2023 Oct;11(5):e003666. doi: 10.1136/bmjdrc-2023-003666. PMID 37797963
- [Background] Wolfsdorf JI, Ratner RE. SGLT Inhibitors for Type 1 Diabetes: Proceed With Extreme Caution. Diabetes Care. 2019 Jun;42(6):991-993. doi: 10.2337/dci19-0008. No abstract available. PMID 31110116
- [Background] Ramphul K, Joynauth J. An Update on the Incidence and Burden of Diabetic Ketoacidosis in the U.S. Diabetes Care. 2020 Dec;43(12):e196-e197. doi: 10.2337/dc20-1258. Epub 2020 Oct 13. No abstract available. PMID 33051332
- [Background] Charleer S, Mathieu C, Nobels F, De Block C, Radermecker RP, Hermans MP, Taes Y, Vercammen C, T'Sjoen G, Crenier L, Fieuws S, Keymeulen B, Gillard P; RESCUE Trial Investigators. Effect of Continuous Glucose Monitoring on Glycemic Control, Acute Admissions, and Quality of Life: A Real-World Study. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1224-1232. doi: 10.1210/jc.2017-02498. PMID 29342264
- [Background] Yau K, Dharia A, Alrowiyti I, Cherney DZI. Prescribing SGLT2 Inhibitors in Patients With CKD: Expanding Indications and Practical Considerations. Kidney Int Rep. 2022 May 5;7(7):1463-1476. doi: 10.1016/j.ekir.2022.04.094. eCollection 2022 Jul. PMID 35812300
- [Background] Simonson GD, Criego AB, Battelino T, Carlson AL, Choudhary P, Franc S, Gershenoff D, Grunberger G, Hirsch IB, Isaacs D, Johnson ML, Kerr D, Kruger DF, Mathieu C, Martens TW, Nimri R, Oser SM, Peters AL, Weinstock RS, Wright EE, Wysham CH, Bergenstal RM. Expert Panel Recommendations for a Standardized Ambulatory Glucose Profile Report for Connected Insulin Pens. Diabetes Technol Ther. 2024 Nov;26(11):814-822. doi: 10.1089/dia.2024.0107. Epub 2024 Jun 10. PMID 38758213
- [Background] Mullen DM, Bergenstal R, Criego A, Arnold KC, Goland R, Richter S. Time Savings Using a Standardized Glucose Reporting System and Ambulatory Glucose Profile. J Diabetes Sci Technol. 2018 May;12(3):614-621. doi: 10.1177/1932296817740592. Epub 2017 Nov 24. PMID 29169243
- [Background] Bergenstal RM, Ahmann AJ, Bailey T, Beck RW, Bissen J, Buckingham B, Deeb L, Dolin RH, Garg SK, Goland R, Hirsch IB, Klonoff DC, Kruger DF, Matfin G, Mazze RS, Olson BA, Parkin C, Peters A, Powers MA, Rodriguez H, Southerland P, Strock ES, Tamborlane W, Wesley DM. Recommendations for standardizing glucose reporting and analysis to optimize clinical decision making in diabetes: the ambulatory glucose profile. J Diabetes Sci Technol. 2013 Mar 1;7(2):562-78. doi: 10.1177/193229681300700234. PMID 23567014
- [Background] Bergenstal RM. Roadmap to the Effective Use of Continuous Glucose Monitoring: Innovation, Investigation, and Implementation. Diabetes Spectr. 2023 Fall;36(4):327-336. doi: 10.2337/dsi23-0005. Epub 2023 Nov 15. PMID 37982061
- [Background] Beck RW, Bergenstal RM, Cheng P, Kollman C, Carlson AL, Johnson ML, Rodbard D. The Relationships Between Time in Range, Hyperglycemia Metrics, and HbA1c. J Diabetes Sci Technol. 2019 Jul;13(4):614-626. doi: 10.1177/1932296818822496. Epub 2019 Jan 13. PMID 30636519
- [Background] Bergenstal RM, Bode BW, Bhargava A, Wang Q, Knights AW, Chang AM. Assessing Time in Range with Postprandial Glucose-Focused Titration of Ultra Rapid Lispro (URLi) in People with Type 1 Diabetes. Diabetes Ther. 2023 Nov;14(11):1933-1945. doi: 10.1007/s13300-023-01476-4. Epub 2023 Sep 23. PMID 37740871
- [Background] Bergenstal RM, Mullen DM, Strock E, Johnson ML, Xi MX. Randomized comparison of self-monitored blood glucose (BGM) versus continuous glucose monitoring (CGM) data to optimize glucose control in type 2 diabetes. J Diabetes Complications. 2022 Mar;36(3):108106. doi: 10.1016/j.jdiacomp.2021.108106. Epub 2021 Dec 31. PMID 35131155
- [Background] Zhang JY, Shang T, Koliwad SK, Klonoff DC. Continuous Ketone Monitoring: A New Paradigm for Physiologic Monitoring. J Diabetes Sci Technol. 2021 Jul;15(4):775-780. doi: 10.1177/19322968211009860. Epub 2021 Apr 9. PMID 33834884
- [Background] Bergenstal RM, Simonson GD, Heinemann L. More Green, Less Red: How Color Standardization May Facilitate Effective Use of CGM Data. J Diabetes Sci Technol. 2022 Jan;16(1):3-6. doi: 10.1177/19322968211053341. Epub 2021 Oct 28. No abstract available. PMID 34711063
- [Background] Tecce N, de Alteriis G, de Alteriis G, Verde L, Tecce MF, Colao A, Muscogiuri G. Harnessing the Synergy of SGLT2 Inhibitors and Continuous Ketone Monitoring (CKM) in Managing Heart Failure among Patients with Type 1 Diabetes. Healthcare (Basel). 2024 Mar 29;12(7):753. doi: 10.3390/healthcare12070753. PMID 38610175
- [Background] Virdi N, Poon Y, Abaniel R, Bergenstal RM. Prevalence, Cost, and Burden of Diabetic Ketoacidosis. Diabetes Technol Ther. 2023 Jun;25(S3):S75-S84. doi: 10.1089/dia.2023.0149. PMID 37306442
- [Background] Danne T, Garg S, Peters AL, Buse JB, Mathieu C, Pettus JH, Alexander CM, Battelino T, Ampudia-Blasco FJ, Bode BW, Cariou B, Close KL, Dandona P, Dutta S, Ferrannini E, Fourlanos S, Grunberger G, Heller SR, Henry RR, Kurian MJ, Kushner JA, Oron T, Parkin CG, Pieber TR, Rodbard HW, Schatz D, Skyler JS, Tamborlane WV, Yokote K, Phillip M. International Consensus on Risk Management of Diabetic Ketoacidosis in Patients With Type 1 Diabetes Treated With Sodium-Glucose Cotransporter (SGLT) Inhibitors. Diabetes Care. 2019 Jun;42(6):1147-1154. doi: 10.2337/dc18-2316. Epub 2019 Feb 6. PMID 30728224
- [Background] Garg SK, Henry RR, Banks P, Buse JB, Davies MJ, Fulcher GR, Pozzilli P, Gesty-Palmer D, Lapuerta P, Simo R, Danne T, McGuire DK, Kushner JA, Peters A, Strumph P. Effects of Sotagliflozin Added to Insulin in Patients with Type 1 Diabetes. N Engl J Med. 2017 Dec 14;377(24):2337-2348. doi: 10.1056/NEJMoa1708337. Epub 2017 Sep 13. PMID 28899222
- [Background] Buse JB, Garg SK, Rosenstock J, Bailey TS, Banks P, Bode BW, Danne T, Kushner JA, Lane WS, Lapuerta P, McGuire DK, Peters AL, Reed J, Sawhney S, Strumph P. Sotagliflozin in Combination With Optimized Insulin Therapy in Adults With Type 1 Diabetes: The North American inTandem1 Study. Diabetes Care. 2018 Sep;41(9):1970-1980. doi: 10.2337/dc18-0343. Epub 2018 Jun 24. PMID 29937430
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Background] Bailey CJ, Day C, Bellary S. Renal Protection with SGLT2 Inhibitors: Effects in Acute and Chronic Kidney Disease. Curr Diab Rep. 2022 Jan;22(1):39-52. doi: 10.1007/s11892-021-01442-z. Epub 2022 Feb 3. PMID 35113333
- [Background] Clegg LE, Heerspink HJL, Penland RC, Tang W, Boulton DW, Bachina S, Fox RD, Fenici P, Thuresson M, Mentz RJ, Hernandez AF, Holman RR. Reduction of Cardiovascular Risk and Improved Estimated Glomerular Filtration Rate by SGLT2 Inhibitors, Including Dapagliflozin, Is Consistent Across the Class: An Analysis of the Placebo Arm of EXSCEL. Diabetes Care. 2019 Feb;42(2):318-326. doi: 10.2337/dc18-1871. Epub 2018 Dec 6. PMID 30523029
- [Background] Menne J, Dumann E, Haller H, Schmidt BMW. Acute kidney injury and adverse renal events in patients receiving SGLT2-inhibitors: A systematic review and meta-analysis. PLoS Med. 2019 Dec 9;16(12):e1002983. doi: 10.1371/journal.pmed.1002983. eCollection 2019 Dec. PMID 31815931
- [Background] Heerspink HJ, Perkins BA, Fitchett DH, Husain M, Cherney DZ. Sodium Glucose Cotransporter 2 Inhibitors in the Treatment of Diabetes Mellitus: Cardiovascular and Kidney Effects, Potential Mechanisms, and Clinical Applications. Circulation. 2016 Sep 6;134(10):752-72. doi: 10.1161/CIRCULATIONAHA.116.021887. Epub 2016 Jul 28. PMID 27470878
- [Background] Neal B, Perkovic V, Matthews DR. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Nov 23;377(21):2099. doi: 10.1056/NEJMc1712572. No abstract available. PMID 29166232